CLINICAL TRIAL: NCT02493231
Title: Effect of Intraoperative Nefopam on Acute Pain After Remifentanil Based Anesthesia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hallym University Kangnam Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, Lee Mi Hyeon, assistant professor, Hallym University Kangnam Sacred Heart Hospital
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: 2014-10-133
Record Dates: First submitted 2015-07-02; First posted 2015-07-09 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-08

CONDITIONS: Cholecystitis
MeSH Terms: conditions — Cholecystitis | interventions — Nefopam; Ketamine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (3):
- Nefopam (Active Comparator): The generic name is 'ACUPAN'. It is infused during operation. A induction dose is 0.3mg/Kg. A maintenance dose is 65 mcg/kg/hr
  Interventions: Drug: Nefopam
- Ketamine (Active Comparator): It is infused during operation. A induction dose is 0.3 mg/Kg. A maintenance dose is 3 mcg/kg/hr
  Interventions: Drug: Ketamine
- Saline (Placebo Comparator): It is infused during operation. A induction volume is 3mL A maintenance dose is 10mL/hr
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Nefopam
  Arms: Nefopam
Drug: Ketamine
  Arms: Ketamine
Drug: Saline
  Arms: Saline

SUMMARY:
Many anesthesiologists use the Remifentanil for reducing a surgical pain and stabilizing a vital sign. However, this drug induce postoperative hyperalgesia. Nowadays, many studies report that low-dose Ketamine prevents the opioid-induces hyperalgesia. Nefopam,which is non-opioid analgesic, has similar mechanism with Ketamine. It will be helpful for postoperative pain control, and reduce the needs of opioid.

ELIGIBILITY:
Inclusion Criteria:

* patient who scheduled laparoscopic cholecystectomy under general anesthesia
* American Society of Anesthesiologist(ASA) class I or II
* adult patient (age 20 - 65)

Exclusion Criteria:

* patient who has liver disease
* patient who has kidney disease
* patient who has diabetes mellitus(DM) or heart disease
* patient who takes opioid or beta-blocker
* patient who has airway disease
* patient who has allergy with the drug

Ages: 20 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-03; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
analgesic requirement | During 1 hour at PACU
duration of analgesic free | During 1 hour at PACU

SECONDARY OUTCOMES:
analgesic requirement | During 8 hours after arriving at ward
Pain on the VAS scale | During 1 hour at PACU

CONTACTS AND LOCATIONS:
Locations (1):
- Hallym University Kangnam Sacred Heart Hospita, Seoul, South Korea